CLINICAL TRIAL: NCT02995096
Title: The Effect of Tumor Characteristics, Pre-transplant Treatments and Immunosuppression on Survival After Liver Transplantation for Hepatocellular Carcinoma - a European Registry Study
Brief Title: Tumor Characteristics, Pre-transplant Treatments and Immunosuppression After Liver Transplantation for Hepatocellular Carcinoma
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Hans-Christian Pommergaard, MD, PhD, Resident, Rigshospitalet, Denmark
Other Study IDs: There is no unique protocol ID
Record Dates: First submitted 2016-12-14; First posted 2016-12-16 (Estimated); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Liver Transplantation
MeSH Terms: interventions — Treatment Expectations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Pre-treatment — Non-transplantation pre-treatments prior to transplantation (e.g. radiofrequency ablation, transcatheter arterial chemoembolization)
Drug: Sirolimus based immunosuppression — Immunosuppression regimens containing Sirolimus

SUMMARY:
Recurrence after liver transplantation for hepatocellular carcinoma (HCC) represents an important cause of mortality for this surgical population. In addition to tumor characteristics, It has been suggested that pre-treatment and sirolimus-based immunosuppression may affect recurrence and survival. With data from the European Liver Transplant Registry (ELTR) database, the aim of this study is to investigate the impact of tumor characteristics, pre-transplant treatment and immunosuppression regimens on survival after liver transplantation for HCC.

ELIGIBILITY:
Inclusion Criteria:

* Hepatocellular carcinoma within transplantation criteria

Exclusion Criteria:

* Disseminated disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients receiving liver transplantation for hepatocellular carcinoma in European centers reporting to the ELTR database.
Sampling Method: Non-Probability Sample
Enrollment: 23124 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Overall survival | up to 10 year survival

SECONDARY OUTCOMES:
Hepatocellular carcinoma specific survival | 5 year and 10 year survival

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Christian Pommergaard, MD, PhD, Principal Investigator — Dept. of Surgery and Transplantion, Rigshospitalet, Denmark

IPD SHARING:
Plan to Share IPD: No
The database material is available for researcher applying for data